CLINICAL TRIAL: NCT02979340
Title: Analysis of Prediction by Ultrasound of the Risk of Hepatic Cirrhosis in Cystic Fibrosis (PUSH) Cohort Using Advanced MRI to Characterize and Predict CF Liver Disease
Brief Title: MRI to Characterize and Predict CF Liver Disease in PUSH Cohort
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CFLD-MRE; U01DK062456 (NIH)
Record Dates: First submitted 2016-11-18; First posted 2016-12-01 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis Liver Disease; Pancreatic Insufficiency
Keywords: Cystic Fibrosis Liver Disease; Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MRI — non-invasive assessment of hepatic fibrosis and steatosis

SUMMARY:
Specific Aim 1. Determine if valid results of non-sedated MRI based assessments of liver stiffness and lipid content can be obtained in more than 90% of children and young adults with cystic fibrosis.

Specific Aim 2. Determine hepatic lipid content using the HepaFat sequence and liver stiffness using MRE. Investigators will compare the results obtained by MRI with PUSH study grayscale ultrasounds in CF patients with normal, heterogeneous, homogeneous or nodular (cirrhotic) pattern on ultrasound.

Specific Aim 3. Creation of an imaging core lab to centralize evaluation of MR imaging data, allow for remote image upload, electronic data storage, and remote image viewing/interpretation. This infrastructure will be utilized to standardize image post processing.

Specific Aim 4. Using the longitudinal PUSH study, determine if MRI based imaging improves discrimination of subjects at risk for progression to advanced CF liver disease (development of cirrhosis) compared to using US imaging alone

DETAILED DESCRIPTION:
This proposal will be a cross sectional study of the current well-characterized PUSH cohort. Patients will receive an MRI at the time of their scheduled PUSH ultrasound. Ideally, the MRI will be performed the same day or a similar time point near liver ultrasound (+/-90 days, but Investigators will allow a larger window due to the slow progression of fibrosis).

Blinded radiology review of imaging sequences will be performed by a local study radiologist with central review performed by the Imaging Core. Analysis by the Imaging Core will include calculation of the liver stiffness, liver and spleen volume, and hepatic and lipid content for all MRI studies.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in longitudinal follow up in PUSH study at a site with MR elastography.

Exclusion Criteria:

1. Age under 6 years (all current patients at time of opening of this study will be greater than 6 years of age).
2. Internal appliance or hardware that is not compatible with MR.
3. Inability to obtain MRI within 6 months of US.
4. Inability to cooperate with MRI.

Ages: 6 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 3 through 12 years of age at time of enrollment diagnosed with Cystic Fibrosis and pancreatic insufficiency and enrolled in the CFLD PUSH longitudinal study.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Change over Time in Liver stiffness and Lipid content over time using MRE | BSL, Year 1, Year 2
  Analysis of variance (ANOVA) will be used to compare the distribution of liver stiffness (in kPa) and lipid content measures between all groups defined by PUSH study grayscale ultrasounds results over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Towbin AJ, Ye W, Huang S, Karmazyn BW, Molleston JP, Masand P, Leung DH, Chang S, Narkewicz MR, Alazraki AL, Freeman AJ, Otto RK, Green N, Kamel IR, Karnsakul WW, Magee JC, Tkach J, Palermo JJ. Prospective study of quantitative liver MRI in cystic fibrosis: feasibility and comparison to PUSH cohort ultrasound. Pediatr Radiol. 2023 Oct;53(11):2210-2220. doi: 10.1007/s00247-023-05706-6. Epub 2023 Jul 28. PMID 37500799
- See also: MRE is a study in the ChiLDReN Network — https://childrennetwork.org